CLINICAL TRIAL: NCT01528930
Title: Inhaled Amikacin for Treatment of Intractable Nontuberculous Mycobacterial Lung Disease
Brief Title: Inhaled Amikacin Treatment for Nontuberculous Mycobacterial Lung Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Although this study was approved at the Institutional Review Board, Korea Food & Drug Administration (KFDA) did not approve this study due to safety concern.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won-Jung Koh, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-104-001
Record Dates: First submitted 2012-01-30; First posted 2012-02-08 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Pulmonary Non-tuberculous Mycobacterial Lung Disease
Keywords: Lung Diseases; Anti-Infective Agents; Therapeutic Uses; Amikacin
MeSH Terms: conditions — Lung Diseases | interventions — Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amikacin for inhalation (Experimental): Drug: Amikacin
  * Amikacin is provided for inhalation via nebulization.
  * 500 mg of amikacin is administered once daily using the Pari-Boy N/Long Life Nebulizer.
  * Administration time is approximately 20 minutes.
  * Amikacin will be administered for 2 years.
  Interventions: Drug: Amikacin

INTERVENTIONS:
Drug: Amikacin — 500 mg, once daily for 2 years

SUMMARY:
The incidence of chronic pulmonary disease caused by nontuberculous mycobacteria (NTM) in human immunodeficiency virus (HIV)-negative patients has been increasing worldwide. In Korea, the common etiologic pathogens for this disease are Mycobacterium avium complex (MAC) and Mycobacterium abscessus. Treating NTM lung diseases can be extremely difficult and may require multiple drugs.

Amikacin is an effective antibiotic for NTM infection. However, intravenous amikacin treatment is limited by its systemic route of administration and a lot of adverse events. Amikacin inhalation treatment could overcome these limitations and also could be effective for treatment of NTM pulmonary disease due to maintaining a high lung concentration. The purpose of this study is to determine whether amikacin inhalation treatment is effective in patients with MAC infection who experienced treatment failure after standard treatment for more than 6 months or with M. abscessus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NTM lung lung disease in accordance with the 2007 ATS/IDSA criteria.
2. MAC lung disease with persistent sputum culture positive after 6 months of standard treatment
3. M. abscessus lung disease with persistent sputum culture positive after 6 months of standard treatment
4. New case of M. abscessus pulmonary disease after completion of initial 4 weeks intravenous antibiotics treatment

Exclusion Criteria:

1. Subjects with negative sputum culture before starting of this study
2. Forced expiratory volume in 1 second (FEV1) <30% of predicted at screening.
3. Positive in HIV test.
4. Subjects with chronic renal insufficient state (serum creatinine level is more than 2.0 mg/dL)
5. Subjects with decreased liver function (serum total bilirubin level is more than 2 mg/dL or AST or ALT are more than 1.5 times of upper normal limits)
6. Active any malignancy requiring chemotherapy or radiation therapy within one year prior to screening.
7. Subjects with history of allergy to amikacin.
8. Subjects with pregnant state or women of childbearing age with no appropriate contraception.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Culture conversion rates at 6 months | 6 months after starting treatment

SECONDARY OUTCOMES:
Culture conversion rates at 12 months | 12 months after starting treatment
Culture conversion rates at 24 months | 24 months after starting treatment
Assessment of abnormal lab values | For 24 months of treatment
Assessment of adverse events related to the study drug or study device | For 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Won-Jung Koh, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea